CLINICAL TRIAL: NCT03739814
Title: A Phase II Study of Inotuzumab Ozogamicin Followed by Blinatumomab for Ph-Negative CD22-Positive B-Lineage Acute Lymphoblastic Leukemia in Newly Diagnosed Older Adults or Adults With Relapsed or Refractory Disease
Brief Title: Inotuzumab Ozogamicin and Blinatumomab in Treating Patients With Newly Diagnosed, Recurrent, or Refractory CD22-Positive B-Lineage Acute Lymphoblastic Leukemia
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - Awaiting amendment to add new cohort
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-02484; NCI-2018-02484 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A041703 (Other: Alliance for Clinical Trials in Oncology); A041703 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: B Acute Lymphoblastic Leukemia, Philadelphia Chromosome Negative; Recurrent B Acute Lymphoblastic Leukemia; Refractory B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (inotuzumab ozogamicin, blinatumomab) (Experimental): See Detailed Description
  Interventions: Biological: Blinatumomab; Biological: Inotuzumab Ozogamicin
- Cohort 2 (inotuzumab ozogamicin, blinatumomab) (Experimental): See Detailed Description.
  Interventions: Biological: Blinatumomab; Biological: Inotuzumab Ozogamicin

INTERVENTIONS:
Biological: Blinatumomab — Given IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC 544; CMC-544; CMC544; Way 207294; WAY-207294

SUMMARY:
This phase II trial studies how well inotuzumab ozogamicin and blinatumomab work in treating patients with CD22-positive B-lineage acute lymphoblastic leukemia that is newly diagnosed, has come back, or does not respond to treatment. Immunotherapy with monoclonal antibodies, such as inotuzumab ozogamicin and blinatumomab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To confirm tolerability of the combination regimen of inotuzumab ozogamicin followed by blinatumomab.

II. To estimate the 1-year event-free survival of older, transplant-ineligible patients with newly diagnosed, Philadelphia (Ph)-negative, CD22-positive, B-cell acute lymphoblastic leukemia (ALL) treated with inotuzumab ozogamicin induction followed by blinatumomab consolidation. (Cohort 1) III. To estimate the 1-year event-free survival of patients with relapsed or refractory Ph-negative, CD22-positive, B-cell ALL treated with inotuzumab ozogamicin induction followed by blinatumomab consolidation. (Cohort 2)

SECONDARY OBJECTIVES:

I. To estimate the median, 1-year, and 3-year overall survival (OS) in all eligible patients. (Cohort 1) II. To estimate the median, 1-year, and 3-year relapse-free survival (RFS) in all eligible patients. (Cohort 1) III. To estimate the median and 3-year event-free survival (EFS) in all eligible patients. (Cohort 1) IV. To estimate the complete response (CR) rate and overall response rate (ORR, defined as complete response [CR] + complete response with incomplete count recovery [CRi]) to inotuzumab ozogamicin followed by blinatumomab (regimen CR rate and ORR). (Cohort 1) V. To estimate the CR rate and ORR (CR + CRi) to inotuzumab ozogamicin induction alone (induction CR and ORR). (Cohort 1) VI. To estimate the minimal residual disease (MRD) negativity rate in subjects achieving a CR or CRi. (Cohort 1) VII. To estimate the treatment-related mortality with this regimen. (Cohort 1) VIII. To describe the safety and tolerability of this regimen. (Cohort 1) IX. To estimate the median, 1-year, and 3-year OS in all eligible patients. (Cohort 2) X. To estimate the median, 1-year, and 3-year RFS in all eligible patients. (Cohort 2) XI. To estimate the median and 3-year EFS in all eligible patients. (Cohort 2) XII. To estimate ORR (CR/CRi and CR/complete response with partial hematologic recovery [CRh]) to blinatumomab in patients with ALL refractory to inotuzumab ozogamicin. (Cohort 2) XIII. To estimate the CR, CRi, and CRh rates at defined time points and cumulatively for the entire regimen. (Cohort 2) XIV. To determine the MRD negativity (< 10^-4) rate at defined time points including prior to allogeneic HCT and cumulatively in patients achieving a CR, CRh, or CRi. (Cohort 2) XV. To determine the allogeneic hematopoietic cell transplantation (HCT) rate in eligible subjects. (Cohort 2) XVI. To estimate the treatment-related mortality with this regimen. (Cohort 2) XVII. To describe the safety and tolerability of this regimen. (Cohort 2)

OTHER OBJECTIVES:

I. Results of the primary analysis will be examined for consistency, while accounting for the stratification factors and/or covariates of baseline quality of life (QOL) and fatigue.

CORRELATIVE SCIENCE OBJECTIVES:

I. To correlate specific karyotype groups (normal or various primary and secondary chromosomal abnormalities) with clinical and laboratory parameters.

II. To correlate specific karyotype groups with response rates, response duration, survival, and cure in patients treated with inotuzumab ozogamicin followed by blinatumomab.

III. To correlate specific karyotype groups with MRD. IV. To determine karyotype changes at relapse and the influence of the type of change (or no change) in karyotype at relapse.

V. To assess the correlation of quantitative MRD post-induction with inotuzumab ozogamicin and at sequential consolidation time points with blinatumomab with RFS, EFS, and OS.

VI. To correlate the influence of MRD status (detectable versus [vs.] not and as a continuous measure) in relation to EFS, RFS, and OS with other clinical and biological factors (e.g. previously untreated vs. relapsed disease cohorts; age, initial white blood cell [WBC] count, cytogenetics).

VII. To identify genetic variants and predictors of ex vivo resistance. VIII. To identify genetic variants and predictors of MRD. IX. To identify genetic variants and predictors of relapse. X. To determine inter-patient variability in drug sensitivity of adult ALL. XI. To examine the associations of drug sensitivity with host and leukemia molecular features.

EXPLORATORY OBJECTIVES:

I. To estimate the median, 1-year, and 3-year RFS, EFS, and OS in patients achieving a CR/CRi to inotuzumab ozogamicin. (Cohort 1) II. To compare the median, 1-year, and 3-year RFS, EFS, and OS among patients achieving MRD-negative vs. MRD-positive CR/CRi to inotuzumab ozogamicin. (Cohort 1) III. To compare the median, 1-year, and 3-year RFS, EFS, and OS among patients achieving MRD-negative vs. MRD-positive CR/CRi at any time. (Cohort 1) IV. To describe the rate, severity, and timing of sinusoidal obstruction syndrome/veno-occlusive disease (SOS/VOD) of the liver after limited inotuzumab ozogamicin exposure and identify risk factors for SOS/VOD. (Cohort 1) V. To estimate the rate of cytokine release syndrome in this population. (Cohort 1) VI. To estimate the median, 1-year, and 3-year RFS from time of CR/CRi to inotuzumab ozogamicin in patients receiving inotuzumab ozogamicin followed by blinatumomab and not undergoing allogeneic hematopoietic cell transplantation (HCT). (Cohort 2) VII. To estimate median, 1-year, and 3-year OS after CR/CRi to inotuzumab ozogamicin in patients not undergoing allogeneic HCT. (Cohort 2) VIII. To compare in a non-randomized fashion median, 1-year, and 3-year OS, median, 1-year, and 3-year RFS, cumulative incidence of relapse (CIR), and non-relapse mortality (NRM) between patients achieving CR/CRi and receiving consolidation with or without allogeneic HCT. (Cohort 2) IX. To describe the rate, severity, and timing of sinusoidal obstruction syndrome/veno-occlusive disease (SOS/VOD) of the liver after limited inotuzumab ozogamicin exposure and identify risk factors for SOS/VOD. (Cohort 2) X. To estimate the rate of cytokine release syndrome in this population. (Cohort 2)

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT 1: Patients receive inotuzumab ozogamicin intravenously (IV) over 1 hour on day 1, 8, and 15 (Course IA). By the end of Course IA (day 21), patients with adequate ALL cytoreduction continue to Course IB/IC, and patients who fail to achieve ALL cytoreduction continue to Course II. By the end of Course II, patients with CR-CRi to Course IB/IC and Course II continue to Course IIIA, patients without adequate ALL cytoreduction to Course IA or refractory to Course IB/IC but CR/CRi to Course II continue to Course IIIB.

COHORT 2: Patients receive inotuzumab ozogamicin IV over 1 hour on day 1, 8, and 15 (Course IA). By the end of Course IA (day 21), patients with adequate ALL cytoreduction continue to Course IB/IC, and patients who fail to achieve ALL cytoreduction continue to Course II. Patients with CR/CRi at the end of Course II continue to Course IIIB.

COURSE IB/IC: Patients receive inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Treatment continues for 1 course (28 days) in the absence of disease progression or unacceptable toxicity.

COURSE II: Patients receive blinatumomab IV continuously on days 1-28 and 43-70. Treatment continues for 1 course (84 days) in the absence of disease progression or unacceptable toxicity.

COURSE IIIA: Patients receive blinatumomab IV continuously on days 1-28 and 43-70. Treatment continues for 1 course (84 days) in the absence of disease progression or unacceptable toxicity.

COURSE IIIB: Patients receive blinatumomab IV continuously on days 1-28, 43-70, and 85-112. Treatment continues for 1 course (126 days) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years, and then every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Pre-registration Eligibility Criteria (Step 0)
* Submission of bone marrow aspirate and peripheral blood for MRD analysis is mandatory prior to registration; the bone marrow sample should be from the first aspiration (i.e. first pull). Aspirate needle should be redirected if needed to get first pull bone marrow aspirate. It should be initiated as soon as possible after pre-registration. The specimens should be sent to the HEME Biobank.

  * Lumbar Puncture (Spinal Tap) and Intrathecal Methotrexate:

    * Patients may receive the day 1 of course IA dose of intrathecal (IT) methotrexate during the prior-to-registration lumbar puncture (or the venous line placement) to avoid a second lumbar puncture. If the dose is administered prior to registration, then systemic chemotherapy must begin within 7 days of this IT chemotherapy.
* Registration Eligibility Criteria (Step 1)
* Morphologic diagnosis of precursor B-cell acute lymphoblastic leukemia (ALL) based on World Health Organization (WHO) criteria. Patients with Burkitt lymphoma/leukemia are not eligible.
* CD22-positive disease defined as CD22 expression by >= 20% of lymphoblasts by local hematopathology evaluation.
* Philadelphia chromosome/BCR-ABL1-negative ALL by cytogenetics, fluorescence in situ hybridization (FISH), and/or polymerase chain reaction (PCR). If any test is positive for Philadelphia chromosome/BCR-ABL1, then the patient is ineligible.
* No active central nervous system (CNS) leukemia (i.e. only CNS-1 disease allowed). Active CNS leukemia is defined as morphologic evidence of lymphoblasts in the cerebrospinal fluid (CSF), use of CNS-directed local treatment for active disease within 28 days prior to registration, symptomatic CNS leukemia (i.e. cranial nerve palsies or other significant neurological dysfunction) within the 28 days prior to registration, and/or known asymptomatic parenchymal CNS mass lesions; see below for additional guidance. Prophylactic intrathecal medication alone is not an exclusion.

  * Categories of CNS Involvement for CNS Evaluation Prior to Registration:

    * CNS 1: CSF has < 5 WBC/uL with cytospin negative for blasts; or >= 10 red blood cell (RBC)/uL with cytospin negative for blasts.
    * CNS 2: CSF has < 5 WBC/uL with cytospin positive for blasts; or >= 10 RBC/uL with cytospin positive for blasts; or >= 10 RBC/uL, WBC/uL >= 5 but less than Steinherz/Bleyer algorithm with cytospin positive for blasts (see below).
    * CNS 3: CSF has >= 5 WBC/uL with cytospin positive for blasts; or >= 10 RBC/uL, >= 5 WBC/uL and positive by Steinherz/Bleyer algorithm (see below); or clinical signs of CNS leukemia (such as facial nerve palsy, brain/eye involvement or hypothalamic syndrome). Steinherz/Bleyer Method of Evaluating Initial Traumatic Lumbar Punctures:

      * If the patient has leukemia cells in the peripheral blood and the lumbar puncture is traumatic and contains >= 5 WBC/uL with blasts, the following algorithm should be used to define CNS disease: CSF WBC/CSF RBC > 2 x (Blood WBC/Blood RBC count)
* Patients with known or suspected testicular involvement by leukemia are allowed provided that the patient receives concomitant scrotal/testicular radiotherapy.

  * Unilateral or bilateral testicular enlargement should be assessed by ultrasound or other imaging technique. Biopsy is recommended if clinical findings are equivocal or suggestive of hydrocele or a non-leukemic mass, but further assessments are per treating physician discretion.
* Not pregnant and not nursing.

  * This study involves agents that have known genotoxic, mutagenic, and teratogenic effects. Therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required.
* Eastern Cooperative Oncology Group (ECOG) performance status: 0-2
* No unstable cardiac disease such as myocardial infarction, angina pectoris, uncontrolled heart failure, or uncontrolled cardiac arrhythmia within 6 months of registration.
* No impaired cardiac function, defined as left ventricular ejection fraction (LVEF) < 45% or New York Heart Association (NYHA) stage III or IV congestive heart failure (CHF).
* Patients with known human immunodeficiency virus (HIV) infection are eligible if they have been on effective antiretroviral therapy with an undetectable viral load tested within 6 months of registration.
* Patients with hepatitis B virus (HBV) are eligible only if they meet all the following:

  * On HBV-suppressive therapy.
  * No evidence of active virus.
  * No evidence of HBV-related liver damage.
* Patients with hepatitis C virus (HCV) are eligible only if they meet all the following:

  * Successfully completed complete-eradication therapy with undetectable viral load.
  * No evidence of HCV-related liver damage.
* No history of clinically relevant neurologic disorder such as epilepsy, seizure, aphasia, stroke, severe brain injury, structural brain abnormality, benign brain tumor, dementia, Parkinson's disease, movement disorder, cerebellar disease, or other significant CNS abnormalities.
* No prior additional malignancy (i.e. in addition to ALL) except adequately treated basal- or squamous-cell skin cancer, in situ cervical cancer, stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for >= 2 years.
* No history of clinically significant ventricular arrhythmia, unexplained non-vasovagal syncope, or chronic bradycardic states such as sinoatrial block or higher degree of atrioventricular block unless a permanent pacemaker has been implanted.
* No history of chronic liver disease, including cirrhosis.
* No history of sinusoidal occlusion syndrome/veno-occlusive disease of the liver.
* No uncontrolled infection or recent history (within 4 months prior to registration) of deep tissue infections such as fasciitis or osteomyelitis.
* Total bilirubin, serum =< 1.5 x upper limit of normal (ULN)*

  * Except in the event of: 1) Gilbert disease, in which case total bilirubin must be =< 2 x ULN, or 2) elevated bilirubin believed by investigator to be due to leukemic infiltration, in which case total bilirubin must be =< 2 x ULN.
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine, serum =< 1.5 ULN OR creatinine clearance >= 40 mL/min
* QT interval by Fridericia's correction formula (QTcF) =< 470 msec
* Cohort 1 Patients Only
* Age >= 60 years.
* No prior treatment for ALL except a single dose of intrathecal chemotherapy, corticosteroids, hydroxyurea, and/or leukapheresis to reduce peripheral blast count and prevent ALL complications. Allowed therapy may be administered for no more than 14 days and must be completed >= 24 hours prior to the initiation of protocol therapy.
* No plan for allogeneic or autologous hematopoietic cell transplantation (HCT).
* Cohort 2 Patients Only:
* Age >= 18 years.
* Relapsed or refractory disease in salvage 1 or 2.
* No isolated extramedullary relapse.
* Prior allogeneic HCT permitted.
* Patients with prior allogeneic HCT must have completed transplantation >= 4 months prior to registration.
* Patients with prior allogeneic HCT must have no evidence of graft-versus-host disease and must have completed immunosuppressive therapy >= 30 days prior to registration.
* Prior treatment with inotuzumab ozogamicin, blinatumomab, other CD22-directed therapy, or other CD19-directed therapy is not allowed.
* Prior treatment with rituximab must be completed >= 7 days prior to registration.
* Prior treatment with other monoclonal antibodies must be completed >= 6 weeks prior to registration.
* Prior treatment for ALL must be completed >= 14 days prior to registration with the following exceptions: intrathecal chemotherapy, hydroxyurea, corticosteroids, 6-mercaptopurine, methotrexate, vincristine, and/or leukapheresis to reduce circulating absolute lymphoblast count to =< 10,000/uL or prevent complications related to ALL are allowed but must be completed >= 24 hours prior to the initiation of protocol therapy.
* Patients should have resolution of any acute non-hematologic toxicities of prior therapy to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 grade =< 1.
* Peripheral blood absolute lymphoblast count =< 10,000/uL (treatment allowed as above to reduce blast count to =< 10,000/uL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | At 1 year
  Will be defined as time from start of treatment to failure to achieve complete response (CR)/complete response with incomplete count recovery (CRi) after completing Course II of blinatumomab, relapse after CR/CRi, progression on study requiring withdrawal from study therapy, or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | Time from start of study therapy to death from any cause censored at the last known alive date, assessed up to 10 years
  Will be evaluated using the Kaplan-Meier method. A 95% confidence interval for the 1- and 3-year rates will be constructed using a point-wise confidence interval for the survival function based on a log-minus-log transformation. Will also calculate a 95% confidence interval by using a point-wise confidence interval for the survival function based on a log-minus-log transformation.
Relapse-free survival (RFS) | Time from first CR/CRi to progressive disease (relapse, treatment discontinuation due to health deterioration) or death, assessed up to 10 years
  Will be evaluated using the Kaplan-Meier method. A 95% confidence interval for the 1- and 3-year rates will be constructed using a point-wise confidence interval for the survival function based on a log-minus-log transformation. Will also calculate a 95% confidence interval by using a point-wise confidence interval for the survival function based on a log-minus-log transformation.
Event-free survival (EFS) | Time from start of treatment to failure to achieve CR/CRi after completing Course II of blinatumomab, relapse after CR/CRi, progression on study requiring withdrawal from study therapy, or death from any cause, assessed up to 10 years
  Will be evaluated using the Kaplan-Meier method. A 95% confidence interval for the 1- and 3-year rates will be constructed using a point-wise confidence interval for the survival function based on a log-minus-log transformation. Will also calculate a 95% confidence interval by using a point-wise confidence interval for the survival function based on a log-minus-log transformation.
Complete and overall response rate | Up to 10 years
  Point and interval estimates of the rates will be shown using a 95% binomial confidence interval.
Minimal residual disease negativity | Up to 10 years
Allogeneic hematopoietic cell transplantation rate (Cohort 2) | Up to 10 years
  Point and interval estimates of the rate will be shown using a 95% binomial confidence interval.

OTHER OUTCOMES:
Rate of cytokine release syndrome (Cohort 1) | Up to 10 years
  Point and interval estimates of the rate will be shown using a 95% binomial confidence interval.
Sinusoidal obstruction syndrome/veno-occlusive disease (SOS/VOD) of the liver | Up to 10 years
  The rate of, timing of, and risk factors for SOS/VOD of the liver after limited inotuzumab ozogamicin exposure. Point and interval estimates of the rate will be shown using a 95% binomial confidence interval. A summary of the timing and risk factors for SOS/VOD of the liver will be provided.
OS | Up to 2 years
  Will compare between patients achieving CR/CRi and receiving consolidation with allogeneic hematopoietic cell transplantation versus (vs.) patients achieving CR/CRi and receiving consolidation without allogeneic hematopoietic cell transplantation. The median, 1-year, and 2-year OS will be compared between the above two groups. The distribution of OS for each group will be estimated using the Kaplan-Meier method.
RFS | Up to 2 years
  Will compare between patients achieving CR/CRi and receiving consolidation with allogeneic hematopoietic cell transplantation vs. patients achieving CR/CRi and receiving consolidation without allogeneic hematopoietic cell transplantation. The median, 1-year, and 2-year RFS will be compared between the above two groups. The distribution of RFS for each treatment arm will be estimated using the Kaplan-Meier method.
Cumulative incidence of relapse (CIR) | Up to 2 years
  Will compare between patients achieving CR/CRi and receiving consolidation with allogeneic hematopoietic cell transplantation vs. patients achieving CR/CRi and receiving consolidation without allogeneic hematopoietic cell transplantation. Competing risk analysis will be done to compare the relapse rates between the above two groups. In this analysis, death will be considered a competing event. Relapse rates at the 1-year and 2-year time points will be estimated. Other time points of interest may be estimated as well.
Non-relapse mortality | Up to 2 years
  Will compare between patients achieving CR/CRi and receiving consolidation with allogeneic hematopoietic cell transplantation vs. patients achieving CR/CRi and receiving consolidation without allogeneic hematopoietic cell transplantation. Competing risk analysis will be done to compare the mortality rates between the above two groups. In this analysis, relapse will be considered a competing event. Mortality rates at the 1-year and 2-year time points will be estimated. Other time points may be estimated as well.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Wieduwilt, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (270):
- United States (270):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Mercy Medical Center, Springfield, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

REFERENCES:
- [Derived] Wieduwilt MJ, Yin J, Kour O, Teske R, Stock W, Escherich C, Yang J, Li Z, Byrd K, Doucette K, Mangan J, Hall S, Mims AS, Jamieson K, Dinner SN, Bseiso AW, Giordano G, Saygin C, Uy GL, Litzow MR, Stone RM. Inotuzumab Ozogamicin Then Blinatumomab for Older Adults With Newly Diagnosed B-Cell ALL: Alliance Study A041703 Cohort 1 Results. J Clin Oncol. 2025 Nov 10;43(32):3526-3535. doi: 10.1200/JCO-25-00307. Epub 2025 Sep 30. PMID 41026957
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074